CLINICAL TRIAL: NCT00636142
Title: A Prospective Trial of Anti-TNF-Alpha Chimeric Monoclonal Antibody (Infliximab, Remicade®) on Insulin Sensitivity, Beta Cell Function and Cardiovascular Risk Profile in Insulin Resistant Human Obesity
Brief Title: Effects of Infliximab on Insulin Sensitivity and Beta Cell Function in Insulin Resistant Human Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Thomas C. Wascher, MD, Department of Internal Medicine, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-000181-39
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Obesity; Insulin Resistance; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Insulin Resistance; Metabolic Syndrome | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Infliximab
  Interventions: Biological: Infliximab
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — 5 mg/kg body weight, maximal dose 500 mg; intravenous administration
  Other Names: Remicade; EU/1/99/116/001-003

SUMMARY:
The aim of the study is to test whether neutralizing TNF-alpha with infliximab affects insulin resistance and phenotypical manifestations of the metabolic syndrome as fasting plasma insulin, total body fat, plasma lipid profile or vascular endothelial function in obese male subjects.

DETAILED DESCRIPTION:
Overweight and obesity are rapidly becoming one of the most pressing health problems. Obese subjects face an increased risk for cardiovascular events that is closely related to a cluster of metabolic disturbances (i.e. insulin resistance, hypertension, dyslipidemia and impaired fibrinolysis), collectively referred to as syndrome X. The actual mechanism underlying development of syndrome X has not been elucidated. Increased TNF-alpha activity has been proposed as a key factor.

The objectives of the study are to test whether neutralizing TNF-alpha with infliximab in obese subjects affects insulin resistance and phenotypical manifestations of the metabolic syndrome such as:

* fasting plasma insulin
* ivGTT derived parameters of insulin resistance and beta-cell function
* total body fat
* plasma lipid profile
* vascular endothelial dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Men, 20-50 years
* BMI 30-35 kg/m2
* HOMA index > 2.5
* stable weight (+/- 2 kg) > 3 months
* Blood pressure>135/85 mmHg (or treated hypertension)
* Triglycerides>1.7 mmol/l or HDL-cholesterol<1.3 mmol/l

Adequate birth control measures for the duration of the study and should continue such precautions for 6 months after receiving the last infusion.

Hemoglobin >= 8.5 g/dL WBC >= 3.5 x 109/L Neutrophils >= 1.5 x 109/L Platelets >= 100 x 109/L SGOT (AST) and AP <3xULN

Chest radiograph within 3 months prior to first infusion with no evidence of malignancy, infection or fibrosis.

No history of latent or active TB prior to screening. No signs or symptoms suggestive of active TB upon medical history and/or physical examination.

No recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study agent.

Within 1 month prior to the first administration of study agent, either have a negative tuberculin skin test or have a newly identified positive tuberculin skin test during screening in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study agent Have a chest radiograph taken within 3 months prior to the first administration of study agent with no evidence of current active TB or old inactive TB.

Exclusion Criteria:

* Overt Diabetes mellitus
* Current treatment with angiotensin II antagonists or ACE inhibitors.
* Treatment indication with statins according to the current NCEP III criteria.
* Treatment indication with low dose acetylsalicylic acid according to the current AHA guidelines or any other NSAID.
* Current smokers.
* Patients with (a history of) an autoimmune disease.
* Use of any investigational drug within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
* Treatment with any other therapeutic agent targeted at reducing TNFα within 3 months of screening.
* Previous administration of infliximab.
* History of receiving human/murine recombinant products or known allergy to murine products.
* Serious infections (such as pneumonia or pyelonephritis) in the previous 3 months. Less serious infections (such as acute upper respiratory tract infection [colds] or simple urinary tract infection) need not be considered exclusions at the discretion of the investigator.
* Documented HIV infection.
* Active hepatitis- B or antibodies against hepatitis-C
* History of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, prior to screening.
* Have or have had a opportunistic infection within 6 months prior to screening.
* Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease (including demyelinating diseases such as multiple sclerosis).
* Concomitant congestive heart failure, including medically controlled asymptomatic patients.
* Presence of a transplanted organ
* Malignancy within the past 5 years.
* History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location or splenomegaly.
* Known recent substance abuse (drug or alcohol).
* Have had a Bacille Calmette-Guerin (BCG) vaccination within 12 months of screening.
* Have a chest radiograph within 3 months prior to randomization that shows an abnormality suggestive of a malignancy or current active infection, including TB.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in fasting insulin levels | 70 days

SECONDARY OUTCOMES:
Blood pressure; Vascular reactivity; Blood measurements + calculation of the HOMA; Iv-GTT; Body fat mass (DEXA); Safety; | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Wascher, MD, Principal Investigator — Medical University of Graz, Graz, Austria
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Wascher TC, Lindeman JH, Sourij H, Kooistra T, Pacini G, Roden M. Chronic TNF-alpha neutralization does not improve insulin resistance or endothelial function in "healthy" men with metabolic syndrome. Mol Med. 2011 Mar-Apr;17(3-4):189-93. doi: 10.2119/molmed.2010.00221. Epub 2010 Nov 16. PMID 21103669